CLINICAL TRIAL: NCT03854019
Title: Evaluating the Efficacy of Dextromethorphan/Quinidine in Treating Irritability in Huntington's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Cures Within Reach (Other)
Responsible Party: Principal Investigator, Erin Furr Stimming, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC-MS-18-1049
Record Dates: First submitted 2019-02-22; First posted 2019-02-26 (Actual); Results first posted 2024-01-05 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Huntington Disease; Irritability
Keywords: Irritability
MeSH Terms: conditions — Huntington Disease | interventions — Dextromethorphan; Quinidine; dextromethorphan - quinidine combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg), then Placebo (Experimental): Dextromethorphan/quinidine (DM/Q) 20mg/10mg one capsule once daily for 1 week, followed by DM/Q 20mg /10 mg twice daily for subsequent 4 weeks, and finally DM/Q 20mg/10mg once daily for 7days.
  Interventions: Drug: Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg); Drug: Placebo
- Placebo, then Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg) (Placebo Comparator): Placebo one capsule once daily for 1 week, followed by placebo twice daily for subsequent 4 weeks, and finally placebo once daily for 7days.
  Interventions: Drug: Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg); Drug: Placebo

INTERVENTIONS:
Drug: Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg) — DM/Q 20mg/10mg one capsule once daily for 1 week, followed by DM/Q 20mg /10 mg twice daily for subsequent 4 weeks, and finally DM/Q 20mg/10mg once daily for 7days.
  Other Names: Nuedexta
Drug: Placebo — Placebo once daily for 1 week, followed by placebo twice daily for subsequent 4 weeks, and finally placebo once daily for 7days.

SUMMARY:
The purpose of this study is to assess efficacy and safety of dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg) in patients with irritability due to Huntington's disease.

ELIGIBILITY:
Inclusion Criteria:

* Verified HD mutation carriers;
* Irritable as diagnosed by the Irritability Scale with a score > 14;
* Stable concomitant medication (no change of medication during last 30 days prior to inclusion);
* Written informed consent by prospective study participant before conduct of any trial-related procedure. Participant must be able to make an informed decision of whether or not to participate in the study.

Exclusion Criteria:

* Hypersensitivity to dextromethorphan (e.g., rash, hives), quinine, mefloquine, quinidine, or dextromethorphan/quinidine with a history of thrombocytopenia, hepatitis, bone marrow depression or lupus-like syndrome induced by these drugs;
* Pregnant or nursing women;
* Active suicidality based on the answer "yes" in questions 4 and 5 of the Columbia-Suicide Severity Rating Scale (baseline version);
* Woman of childbearing potential, not using highly effective methods of contraception such as oral, topical or injected contraception, IUD, contraceptive vaginal ring, or double barrier method such as diaphragm and condom with spermicide) or not surgically sterile (via hysterectomy, ovarectomy or bilateral tubal ligation) or not at least one year post-menopausal;
* Male not using an acceptable barrier method for contraception;
* Presence of any medically not controllable disease (e.g. uncontrolled arterial hypertension or diabetes mellitus);
* Clinically significant renal (calculated creatinine clearance < 30 ml/min) or hepatic dysfunction;
* Patients with pre-existing hepatic disease;
* Individuals with a history or complete heart block, QTc prolongation or tornadoes de pointes, or at high risk of complete AV block;
* Family history of congenital QT prolongation;
* History of unexplained syncope within the past year;
* Use of drugs containing quinidine, quinine, or mefloquine;
* Individuals currently taking strong CYP3A4 inhibitors or tetrabenazine;
* Use of certain antidepressants--amitriptyline, clomipramine, desipramine, fluoxetine, paroxetine, sertraline, venlafaxine;
* Use of certain heart rhythm medications--amiodarone, flecainide, procainamide, propafenone;
* Use of certain medicines to treat psychiatric disorders--chlorpromazine, haloperidol, perphenazine, pimozide, quetiapine, risperidone, thioridazine.
* Use of tamoxifen;
* Presence or history of seizures or diagnosed epilepsy;
* Severe cognitive disorders defined as a score < 18 on the MOCA;
* Clinically relevant abnormal findings in the ECG, the vitals, in the physical examination or laboratory values at screening that could interfere with the objectives of the study or the safety of the subject as judged by the investigator;
* Participation in another investigative drug trial within 2 months;
* Subjects who are unlikely to be compliant and attend scheduled clinic visits as required as determined by the Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-08-05 (Actual); Primary Completion 2022-11-11 (Actual); Study Completion 2022-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erin L Furr Stimming, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zadegan SA, Calderon O, Karagas N, Patino J, Dongarwar D, Duncan B, Teixeira AL, Rocha NP, Furr Stimming E. Assessing the efficacy of dextromethorphan/quinidine in treating irritability in Huntington's disease. J Huntingtons Dis. 2026 Jan 7:18796397251411112. doi: 10.1177/18796397251411112. Online ahead of print. PMID 41499296

RESULTS

PARTICIPANT FLOW:
Period: First Intervention (4 Weeks)
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg), Then Placebo | Placebo, Then Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg)
Started | 10 | 10
Completed | 9 | 9
Not Completed | 1 | 1
Period: Washout (1 Week)
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg), Then Placebo | Placebo, Then Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0
Period: Second Intervention (4 Weeks)
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg), Then Placebo | Placebo, Then Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg)
Started | 9 | 9
Completed | 9 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg), Then Placebo | Placebo, Then Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Total
Number analyzed (Participants) | 9 | 9 | 18
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 9 | 18
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.8 (14.2) | 43.1 (6.3) | 43.9 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 5 | 11
  Male | 3 | 4 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 4 | 7
  Not Hispanic or Latino | 6 | 5 | 11
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 6 | 5 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 4 | 7
Region of Enrollment [Number; unit: participants]
  United States | 9 | 9 | 18

OUTCOME MEASURES:

1. Primary Outcome: Irritability as Assessed by The Irritability Scale.
Description: The Irritability Scale total score ranges from 0 to 42, with higher scores indicating greater irritability.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- All Study Participants Pre-Randomization: All Study Participants Pre-Randomization
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 27.5 (5.8)

2. Primary Outcome: Irritability as Assessed by The Irritability Scale
Description: The Irritability Scale total score ranges from 0 to 42, with higher scores indicating greater irritability.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg): Dextromethorphan/quinidine (DM/Q) 20mg/10mg one capsule once daily for 1 week, followed by DM/Q 20mg /10 mg twice daily for subsequent 4 weeks, and finally DM/Q 20mg/10mg once daily for 7days.
- Placebo: Placebo one capsule once daily for 1 week, followed by placebo twice daily for subsequent 4 weeks, and finally placebo once daily for 7days.
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 18.7 (10.1) | 19.9 (9.4)

3. Secondary Outcome: Behavioral Symptoms, as Assessed by the Hospital Anxiety and Depression Scale (HADS).
Description: The HADS is a self-report, 14-item scale (7 items relate to anxiety and 7 relate to depression) used to determine the levels of anxiety and depression that a person is experiencing. The total score ranges from 0 to 42 (21 per subscale), with higher scores signifying worse symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 16.7 (5.6)

4. Secondary Outcome: Behavioral Symptoms, as Assessed by the Hospital Anxiety and Depression Scale (HADS).
Description: as for outcome 3
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 10.6 (6.7) | 11.1 (8.3)

5. Secondary Outcome: Behavioral Symptoms, as Assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) - Severity Score.
Description: The NPI-Q is a 12-domain informant-based interview that assesses neuropsychiatric symptoms over the previous month.The total NPI-Q severity score ranges from 0 to 36, with higher scores indicate greater symptoms severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 10.4 (4.2)

6. Secondary Outcome: Behavioral Symptoms, as Assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) - Severity Score.
Description: as for outcome 5
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 8.2 (4.5) | 8.6 (6.2)

7. Secondary Outcome: Behavioral Symptoms, as Assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) - Caregiver Distress.
Description: Caregiver distress associated with the symptom is rated on an anchored 0- to 5-point scale, which total sum ranges from 0 to 60. Higher scores indicate greater caregiver distress related to patient's neuropsychiatric symptoms.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 13.1 (6.5)

8. Secondary Outcome: Behavioral Symptoms, as Assessed by the Neuropsychiatric Inventory-Questionnaire (NPI-Q) - Caregiver Distress.
Description: as for outcome 7
Time Frame: 4 weeks
Population: Data were not collected for 1 participant in the Dextromethorphan/quinidine 20mg/10mg (DM/Q 20mg/10mg) arm. Data were not collected for 1 participant in the Placebo arm
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 17 | 17
score on a scale | 7.8 (5.2) | 11.3 (7.4)

9. Secondary Outcome: Behavioral Symptoms, as Assessed by the Problem Behaviors Assessment - Short Version (PBA-s). - Irritability/Aggression Subscale
Description: The PBA-s is a semistructured interview to measure severity and frequency of behavioral problems in Huntington's disease. The PBA-s is an 11-item scale rating the frequency and severity of symptoms. The total score for irritability/aggression subscale ranges from 0 to 32, with higher scores indicating greater behavioral symptoms severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 12.9 (7.2)

10. Secondary Outcome: Behavioral Symptoms, as Assessed by the Problem Behaviors Assessment - Short Version (PBA-s) - Irritability/Aggression Subscale
Description: as for outcome 9
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 7.6 (5.8) | 8.7 (5.7)

11. Secondary Outcome: Motor Symptoms, as Assessed by the Total Motor Score (TMS) From the UHDRS.
Description: The TMS comprises the motor section of the UHDRS, a 31-item subscale that comprehensively evaluates motor aspects of HD. The overall 31 items are each rated from grade 0 (not affected) to grade 4 (most severely affected), resulting in a range of 0-124 points.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 18.7 (11.8)

12. Secondary Outcome: Motor Symptoms, as Assessed by the Total Motor Score (TMS) From the UHDRS.
Description: as for outcome 11
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 19.3 (11.8) | 18.7 (11.5)

13. Secondary Outcome: Motor Symptoms, as Assessed by the Total Maximal Chorea (TMC).
Description: The TMC comprises 7 of the 31 items in the TMS, which are related to chorea symptoms. The total TMC score ranges from 0 to 28, with higher scores indicating greater chorea severity.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 6.0 (3.8)

14. Secondary Outcome: Motor Symptoms, as Assessed by the Total Maximal Chorea (TMC).
Description: as for outcome 13
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 5.9 (4.3) | 5.2 (4.0)

15. Secondary Outcome: Functional Independence, as Assessed by the UHDRS Total Functional Capacity Scale (TFC).
Description: The TFC lists five stages of Huntington's Disease and five levels of function in the domains of workplace, finances, domestic chores, activities of daily living and requirements for unskilled or skilled care. The total TFC score ranges from 0 to 13, with higher scores signifying better functioning.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 11.3 (1.2)

16. Secondary Outcome: Functional Independence, as Assessed by the UHDRS Total Functional Capacity Scale (TFC).
Description: as for outcome 15
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 11.4 (1.7) | 11.3 (1.8)

17. Secondary Outcome: Number of Participants With Behavioral Suicidal Events, as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation.
Description: The C-SSRS is a suicidal ideation and behavior rating scale with yes/no responses. The first part (Items 1-5) rates an individual's degree of suicidal ideation on a 0-5 scale, ranging from "wish to be dead" to "active suicidal ideation with specific plan and intent and behaviors". The C-SSRS outcomes are categories and have binary responses (yes/no). Suicidal ideation is considered when the patient responds a "yes" answer at any time during treatment to any one of the five suicidal ideation questions (Categories 1-5) on the C-SSRS. The sum of the 5 intensity item scores create a total score (range 0 to 25) to represent the intensity rating (higher scores indicate more severe suicidal ideation).
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
Participants | 0

18. Secondary Outcome: Number of Participants With Behavioral Suicidal Events, as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Ideation
Description: as for outcome 17
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

19. Secondary Outcome: Number of Participants With Behavioral Suicidal Events, as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Behavior.
Description: The questions 6-10 of the C-SSRS are related to suicidal behavior, and the outcome is a simple yes/no response. Suicidal behavior occurs if the patient answers a "yes" at any time during treatment to any one of the five suicidal behavior questions (Categories 6-10) on the C-SSRS.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
Participants | 0

20. Secondary Outcome: Number of Participants With Behavioral Suicidal Events, as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) - Suicidal Behavior.
Description: as for outcome 19
Time Frame: 4 Weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
Participants | 0 | 0

21. Secondary Outcome: Cognitive Symptoms, as Assessed by the The Montreal Cognitive Assessment (MoCA).
Description: The MoCA is a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains with a total possible score of 0 to 30 points; a score of 26 or above is considered normal for the general population.
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
score on a scale | 25.3 (3.0)

22. Secondary Outcome: Cognitive Symptoms, as Assessed by the The Montreal Cognitive Assessment (MoCA).
Description: as for outcome 21
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
score on a scale | 26.2 (2.7) | 26.6 (2.3)

23. Secondary Outcome: Patient Progress and Treatment Response Over Time, as Assessed by the Clinical Global Impressions Severity Scale (CGI-S).
Description: The CGI is a stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication.
Time Frame: Baseline
Measure: Count of Participants; unit: Participants
Arm/Group | All Study Participants Pre-Randomization
Number analyzed (Participants) | 18
Participants
  Normal | 0
  Borderline ill | 0
  Mildly ill | 3
  Moderately ill | 11
  Markedly ill | 3
  Severely ill | 0
  Extremely ill | 0
  Not analyzed | 1

24. Secondary Outcome: Patient Progress and Treatment Response Over Time, as Assessed by the Clinical Global Impressions Severity Scale (CGI-S).
Description: The CGI is a stand-alone assessment of the clinician's view of the patient's global functioning prior to and after initiating a study medication. The CGI is a 3-item observer-rated scale that measures illness severity (CGI-S), global improvement or change (CGI-I) and therapeutic response. The scale ranges from 1-7, with higher scores indicating worse outcomes.
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
Participants
  Normal | 0 | 0
  Borderline ill | 1 | 4
  Mildly ill | 2 | 2
  Moderately ill | 14 | 9
  Markedly ill | 0 | 1
  Severely ill | 0 | 0
  Extremely ill | 0 | 0
  Not analyzed | 1 | 2

25. Secondary Outcome: Patient Progress and Treatment Response Over Time, as Assessed by the Clinical Global Impressions Improvement Scale (CGI-I).
Description: as for outcome 23
Time Frame: 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 18 | 18
Participants
  Very much improved | 1 | 1
  Much improved | 4 | 5
  Minimally improved | 3 | 0
  No change | 8 | 9
  Minimally worse | 1 | 0
  Much worse | 0 | 2
  Very much worse | 0 | 0
  Not analyzed | 1 | 1

26. Secondary Outcome: Cognitive Symptoms, as Assessed by the Unified Huntington's Disease Rating Scale (UHDRS) - Cognitive Domain.
Description: The UHDRS - cognitive function assessment a phonetic verbal fluency test, the Symbol Digit Modalities Test, and the Stroop Interference Test. These tests do not have a predefined score range, but higher scores indicate better cognitive performance.
Time Frame: Baseline
Population: Data were not collected for this outcome measure
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 0 | 0

27. Secondary Outcome: Cognitive Symptoms, as Assessed by the Unified Huntington's Disease Rating Scale (UHDRS) - Cognitive Domain.
Description: as for outcome 26
Time Frame: 4 weeks
Population: Data were not collected for this outcome measure
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 13 weeks
Arm/Group | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 1/20
Other Adverse Events (participants affected / at risk) | 10/20 | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) (N=20) | Placebo (N=20)
Hospitalization for motorcycle accident (General disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dextromethorphan/Quinidine 20mg/10mg (DM/Q 20mg/10mg) (N=20) | Placebo (N=20)
Insomnia (General disorders) | 1 | 1
Headaches (General disorders) | 2 | 0
Diarrhea (Gastrointestinal disorders) | 0 | 1
Fingernail infection (Infections and infestations) | 0 | 1
Nausea (General disorders) | 1 | 0
Dizziness (General disorders) | 1 | 0
Loss weight/decreased appetite (General disorders) | 1 | 0
Increased libido (General disorders) | 1 | 0
Decreased libido (General disorders) | 0 | 1
decline in mood (General disorders) | 0 | 1
Primary care physician (PCP) prescribed medication for high blood pressure (General disorders) | 1 | 0
Increased apathy (General disorders) | 1 | 0
COVID-19 (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-01-28): https://cdn.clinicaltrials.gov/large-docs/19/NCT03854019/Prot_SAP_000.pdf